CLINICAL TRIAL: NCT02542566
Title: Randomised Control Trial Comparing Conservative Rehabilitation and Protected Weight Bearing Versus Accelerated Rehabilitation and Early Weight Bearing Post Microfracture Knee Surgery.
Brief Title: Protected Versus Early Weight Bearing Post Microfracture Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped prematurely due to the lack of eligible participants.
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: version 4 28/08/2014
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2015-09

CONDITIONS: Defect of Articular Cartilage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- early weight bearing (Active Comparator): early weight bearing and accelerated physiotherapy rehabilitation
  Interventions: Procedure: Physiotherapy rehabilitation
- protected weight bearing (Active Comparator): protected weight bearing and conservative physiotherapy rehabilitation.
  Interventions: Procedure: Physiotherapy rehabilitation

INTERVENTIONS:
Procedure: Physiotherapy rehabilitation — Physiotherapy rehabilitation

SUMMARY:
To test using a randomised control trial, whether conservative rehabilitation and protected weight bearing versus early weight bearing and accelerated rehabilitation affects patient outcomes post microfracture surgery of the knee.

DETAILED DESCRIPTION:
To test using a randomised control trial, whether conservative rehabilitation and protected weight bearing versus early weight bearing and accelerated rehabilitation affects patient outcomes post microfracture surgery of the knee.

Current practice in most units is to protect patients from weight bearing prior to entering a conservative physiotherapy rehabilitation program following microfracture surgery of the knee. At our unit we believe that protecting patients from weight bearing post microfracture surgery makes no difference to their outcome and only leads to a longer rehabilitation time and a delayed return to work and sports. Therefore we want to randomise patients who require microfracture surgery of the knee for cartilage defects into 2 post operative rehabilitation groups. One group will be able to weight bear early and will undergo an accelerated rehabilitation program whilst the other will be protected from weight bearing and will undergo a more conservative rehabilitation program. We will then follow patients up over a year and compare outcome data collected at 6 weeks, 3 months, 6 months and 1 year post operatively to see if there was any difference in outcomes between the 2 groups. As secondary outcomes we will also compare the patients in the two groups to see if there is a difference in time taken to return to work and sporting activities

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-60 years. Mechanically stable knee joint at outpatient examination. MRI confirmed grade 3 or 4 non-kissing cartilage defect within the knee. Able to fully understand the process and study and give informed consent to participate.

Able to comply with the physiotherapy rehabilitation and follow up process.

Exclusion Criteria:

* Kissing cartilage defects. Defects deemed too large to undergo microfracture on MRI scan. Clinically unstable knee joint. Patients unable to consent to participation. Under 16 years of age or over 60 years of age. Patients likely to drop out of physiotherapy rehabilitation and study follow up.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Modified Tegner/Lysholm score from questionnaires. | 12 months

SECONDARY OUTCOMES:
Time to return to work. | 12 months
Time to return to sporting activities | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gallacher, Surgeon, Study Director — NHS Healthcare
Locations (1):
- The Robert Jones and Agnes Hunt Orthopaedic Hospital NHS FT, Oswestry, Shropshire, United Kingdom